CLINICAL TRIAL: NCT02062086
Title: Estimation of Muscle Mass in Older Adults Using Deuterated Creatine
Acronym: MM-DC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RC31/13/6911; 2013-A01339-36 (Other: ID-RCB)
Record Dates: First submitted 2014-02-06; First posted 2014-02-13 (Estimated); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Sarcopenia
Keywords: Sarcopenia; Mass muscle; Quality of life
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Population 1 (Other): (Community-dwelling older adults) will participate in the study for approximately 65 days.
  Population 1 will absorb deuterated creatine 30 mg, a non-radioactive, stable isotope of creatine, for the estimation of muscle mass in humans.
  The estimation of muscle mass will be made on 2 separate occasions in the community-dwelling elderly population in order to assess reproducibility of the method when tested approximately 60 days apart.
  Interventions: Dietary Supplement: deuterated creatine 30 mg
- Population 2 (Other): (Hip-fracture patients) will participate in the study for approximately 35 days during their in-hospital period, followed by 30 during their post-discharge period, so for a total period of at least 65 days.
  Population 2 will absorb deuterated creatine 30 mg, a non-radioactive, stable isotope of creatine, for the estimation of muscle mass in humans.
  In the hip fracture population, estimation of muscle mass by the D3 creatine method will be performed on up to 3 separate occasions to assess whether the method is sensitive enough to detect decreases in muscle mass that may occur during the recovery period after hip fracture.
  Interventions: Dietary Supplement: deuterated creatine 30 mg

INTERVENTIONS:
Dietary Supplement: deuterated creatine 30 mg — Study participants will take a single oral dose of deuterated creatine 30 mg in capsule form

SUMMARY:
Current methods for the quantification of muscle mass are indirect, lack precision, and often rely on expensive equipment that only provides limited (indirect) data on whole body muscle mass. Dual energy X ray absorptiometry has emerged as a potential precise measure of lean mass, easy to use in clinical practice and research. However, it assesses an indirect measurement of total-body skeletal muscle mass and its clinical use for determination of changes in muscle mass may be very limited due to instrumentation availability, particularly in field studies, and cost. Moreover, these methods provide estimates of fat free mass that is not skeletal muscle specific, and are influenced by changes in regional or total body water content.

GlaxoSmithKline (GSK) has developed a novel technique using deuterium labeled creatine dilution for the estimation of muscle mass and has begun clinical evaluation of this muscle-measure in healthy young and older adults.

DETAILED DESCRIPTION:
Mobility disability in acute and chronic settings like the Frailty day Hospital or the rehabilitation units make it difficult to assess muscle mass other than the availability of imaging techniques. Often it is impossible to assess muscle mass due to accessibility and cost of actual techniques. Deuterium labeled creatine (contained in capsules to be swallowed) is an easy procedure to assess muscle mass that could avoid the existing difficulties when using imaging techniques. Capsules containing the deuterium labeled creatine will be administered to participants who will autonomously take them. The subsequent assessment of urinary deuterium dilution will provide the estimate of skeletal muscle mass of the individual.

Primary outcome: Assess muscle mass quantity in older adults using the method of deuterium labeled creatine versus the DXA (Dual Energy X-ray Absorptiometry) total lean mass assessment.

ELIGIBILITY:
Inclusion criteria

Population 1: Community-dwelling older adults:

* Community-dwelling at the time of the assessment
* Ambulatory without human assistance at the time of the assessment
* ADL (activity of daily living)equal to 5 or more at the time of the assessment

Population 2: Older adults recovering after hip fracture surgery:

* Age ≥ 65 at the time of the fracture
* Minimal trauma hip fracture (Diagnosis of closed fracture of the proximal femur and no history of a fall from height higher than standing height (e.g. fall from a roof or a ladder); no history of a high impact fracture (e.g. car accident, skiing)
* Unilateral hip fracture
* Surgical repair of hip fracture
* Surgical intervention taking place within 7 days since admission to the acute care unit.
* Living in the community at the time of the fracture
* Anticipated discharge back to the community
* Ambulatory without human assistance prior to the fracture
* ADL (activity of daily living) equal to 5 or more prior to the fracture

Exclusion criteria

Population 1:Community-dwelling elderly:

* Diagnosis of dementia
* Presence of cognitive impairment (assessed during clinical follow-up using standardized cognitive tools such as MMSE (Mini Mental Status Examination) or MOCA (Montreal Cognitive Assessment), during pre-screening period).
* Inability to provide informed consent
* Presence of severe or uncontrolled neurodegenerative disease like Parkinson's disease, amyotrophic lateral sclerosis or multiple sclerosis
* Presence of an underlying muscle disease other than age-associated muscle waste or disuse atrophy.
* History of stroke with residual hemiplegia
* Diagnosis of a severe medical or psychiatric condition making the participant unlikely to understand or comply with study protocol.
* Diagnosis of malignancy done in the 18 months prior the baseline visit.
* Severe renal failure

Population 2: Older adults recovering from hip fracture:

* Pathological hip fracture
* Diagnosis of dementia
* Presence of cognitive impairment (assessed during clinical follow-up using standardized cognitive tools such as MMSE (Mini Mental Status Examination) or MOCA (Montreal Cognitive Assessment), during prescreening period).
* Peri-operative delirium persisting after day 5 of post-operative period.
* Inability to provide informed consent
* Presence of severe or uncontrolled neurodegenerative disease like Parkinson's disease, amyotrophic lateral sclerosis or multiple sclerosis
* Presence of an underlying muscle disease other than age-associated muscle waste or disuse atrophy.
* History of stroke with residual hemiplegia
* Diagnosis of a severe medical or psychiatric condition making the participant unlikely to understand or comply with study protocol.
* Diagnosis of malignancy done in the 18 months prior the baseline visit.
* Severe renal failure

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 33 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Muscle mass quantity | Assess muscle mass quantity in older adults using the method of deuterium labeled creatine versus the DXA total lean mass assessment. Modification of the muscle mass quantity between Day 4 and Day 64
  Study participants will take a single oral dose of deuterated creatine 30 mg in capsule form. Muscle mass quantity will be assessed using D3-creatine technique.

SECONDARY OUTCOMES:
Repeatability of muscle mass estimates | Evaluate the repeatability of muscle mass estimates from deuterium labeled creatine dilution method in community dwelling elderly subjects who meet specific "frailty" criteria. The repeatability will be assessed comparing day 4 and day 64
  The estimation of muscle mass will be made on 2 separate occasions in the community-dwelling elderly population in order to assess reproducibility of the method when tested approximately 60 days apart.
Creatine dilution of the deuterium labeled | Evaluate the deuterium labeled creatine dilution for sensitivity to changes in muscle mass in the hip fracture population during the period after fracture when muscle mass is expected to decline. It will be assessed comparing day 4, day 34 and day 64
  Estimation of muscle mass by the D3 creatine method will be performed on up to 3 separate occasions to assess whether the method is sensitive enough to detect decreases in muscle mass that may occur during the recovery period after hip fracture.
Association of muscle mass with measures of lower extremity function, muscle strength and physical activity. | Examine the association of muscle mass with measures of lower extremity function, muscle strength and physical activity.
  Lower extremity function will be assessed longitudinally in both cohorts using:
  Short Physical Performance Battery (SPPB) and The six minute walk test (6-MWT)
  To measure the physical activity:
  Self-reported physical activity - The Minnesota Leisure Time Physical Activity Questionnaire (MLTPAQ) Accelerometer measurement
  To measure muscle strength:
  Leg extension strength Handgrip strength
Association of measures of muscle mass, muscle strength and levels of physical activity with quality of life assessments | Examine the association of measures of muscle mass, muscle strength and levels of physical activity with quality of life assessments and patient reported outcomes.
  * Quality of life assessed by EuroQol.
  * Sarcopenia Patient Reported Outcome Assessment
  * Self-Reported Function Using these questionnaires and measurements, we will try to find out the link between muscle mass, muscle strength, level of physical activity and quality of life
Feasibility of the method | Evaluate the feasibility of developing a blood based assay using deuterium labeled creatine dilution for the estimation of muscle mass.
  The current method is based on analyses from urine sampling; however, plasma samples will also be drawn in this study to evaluate the feasibility of developing a blood based assay. Blood sampling is much easier than urine assessments, so that in future studies blood sampling would be the assessment of choice if the dosing proofs to be feasible.
Correlation between muscle function and muscle mass | Assess if there exists a correlation between muscle function and muscle mass estimated by D3-Creatine
  The study will also explore if not only measures of muscle mass, but also if muscle function are correlated with urine and blood sampling of D3 creatine.

CONTACTS AND LOCATIONS:
Overall Officials: Gabor Abellan Van Kan, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Gerontopôle - CHU La Grave Casselardit - Serv. de Médecine Interne & de Gérontologie Clinique - 170 av de Casselardit - TSA 40031, Toulouse, France